CLINICAL TRIAL: NCT06052878
Title: Association Between Prenatal Anesthesia Exposure and Neurodevelopmental Outcome : an Ambi-directional Cohort Study
Brief Title: Neurodevelopmental Outcome After Prenatal Anesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CHUCaen
Record Dates: First submitted 2023-06-14; First posted 2023-09-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: Neurodevelopmental Disorders; Child Behavior
Keywords: general anesthesia; regional anesthesia; pregnancy; executive functions; developing brain; neurodevelopment; surgery
MeSH Terms: conditions — Neurodevelopmental Disorders; Child Behavior | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General anesthesia: Children whose mothers underwent general anesthesia for non-obstetric surgery during pregnancy.
  Interventions: Other: Parental telephone interview with standardized parental questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF); Other: Parental questionnaire about their child's cognitive functioning in their daily life and medical history.
- Locoregional anesthesia: Children whose mothers underwent regional anesthesia for non-obstetric surgery during pregnancy.
  Interventions: Other: Parental telephone interview with standardized parental questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF); Other: Parental questionnaire about their child's cognitive functioning in their daily life and medical history.
- Control: Children whose mothers did not undergo any surgical intervention during pregnancy.
  Interventions: Other: Parental telephone interview with standardized parental questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF); Other: Parental questionnaire about their child's cognitive functioning in their daily life and medical history.

INTERVENTIONS:
Other: Parental telephone interview with standardized parental questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF) — The "Behaviour Rating Inventory of Executive Function" (BRIEF) is a parental questionnaire that assesses the executive functions of children aged 5 to 18 years old. It consists of 86 questions grouped into 8 scales: inhibition, flexibility, emotional control, initiation, material organization, working memory, planning/organization, and monitoring. It provides information on a global scale (score) regarding subtle and subclinical changes in various executive functions.
Other: Parental questionnaire about their child's cognitive functioning in their daily life and medical history. — Standardized questionnaire includes : The child's medical history and cognitive functioning (at school, parental home, and during extracurricular activities), home environment, parent's child socioeconomic status and emotional climate.

SUMMARY:
In 2016, the US Food and Drug Administration raised concerns about the potential negative effects of anesthesia exposure on neurodevelopment in children during pregnancy or before the age of three.

The impact of exposure to anesthetic agents on neurodevelopmental outcome however remains debated: clinical studies on the subject do not allow for unequivocal conclusions to be drawn, given their methodological heterogeneity and the numerous confounding environmental factors.

To this date, only two studies have focused on the potential neurodevelopmental effects of general anesthesia during the prenatal period, even though general anesthesia for non-obstetric surgery during pregnancy affects up to 3% of pregnant women.

This observational ambidirectional study would be the first to investigate the potential neurodevelopmental effects of prenatal exposure to anesthesia, whether general or regional, for surgery during pregnancy. It would thus differentiate between the contribution of surgical stress and that of anesthetic agents in any observed modifications.

The aim of the study is:

Are there any subtle modifications of executive functions associated with prenatal exposure to anesthesia during non-obstetric surgery during pregnancy?

To investigate this, parents of the participating children will be asked to complete a standardized parental telephone questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF). This parental questionnaire allows for evaluating children's behaviors related to executive functions.

Researchers will compare the score derived from the "BRIEF" parental questionnaire (BRIEF score) between three groups of children aged from 5 to 12 years old, born between 2011 and 2018 at Caen University Hospital:

* The " General anesthesia " group: children whose mothers underwent general anesthesia for non-obstetric surgery during pregnancy (N: 62).
* The " Locoregional anesthesia " group: children whose mothers underwent regional anesthesia for non-obstetric surgery during pregnancy (N: 31).
* The " Control " group: children whose mothers did not undergo any surgical intervention during pregnancy (N: 62).

The first aim of our study is to investigate the presence of a significant difference in the BRIEF score between the three groups.

The seconds aims are to assess the cognitive functioning of patients in their daily lives (school, parental home, and extracurricular activities).

DETAILED DESCRIPTION:
The study : "Association Between Prenatal Anesthesia Exposure and Neurodevelopmental Outcome : an Ambidirectional Cohort Study" is a single-center, ambidirectional, observational cohort study conducted at the University Hospital Center of Caen (CHU Caen).

Inclusion criteria :

The study groups "General Anesthesia" (GA group) and "Locoregional Anesthesia" (LRA group) are derived from a previous Caen University Hospital cohort, consisting of children whose mothers underwent general or regional anesthesia for non-obstetric surgery during pregnancy.

This previous cohort was established in 2021 for an unpublished research project consisting of 179 patients who underwent non-obstetric surgeries during pregnancy. These pregnant women who underwent surgery were identified through the Caen University hospital electronic database spanning from 2011 to 2020, as surgical procedures for pregnant women started to be documented since 2011 in the medical database of this hospital.

The "control group" will be formed by including children born at Caen University Hospital, the same day, right before and right after the children in the LRA group, but whose mothers did not undergo any surgical intervention during pregnancy.

The number of exposed patients (N=93) is comparable to prospective studies investigating the effect of postnatal general anesthesia on neurodevelopmental outcomes. It is also comparable to and higher than the two studies investigating the effect of prenatal general anesthesia on neurodevelopmental outcomes.

Matching :

The matching of the GA and LRA groups will be done based on the following three adjustment factors:

* Socio-economic level (parental monthly net income within a range of 500 euros)
* Age at the time of testing
* Gender of the child

Inclusion process:

After providing the information sheet and receiving the signed consent form from the legal guardian of the child, the elements of the parental telephone interview will be collected from the child's parents, prospectively, on a standardized data collection sheet during an estimated phone call duration of approximately forty minutes.

The phone call will consist of two parts :

* The standardized parental questionnaire from the "Behaviour Rating Inventory of Executive Function" (BRIEF).
* The parental hetero-questionnaire about their child's cognitive functioning in their daily life and medical history.

Both the parental standardized BRIEF questionnaire and our parental hetero-questionnaire will contribute to fulfilling the study objectives.

The parental hetero-questionnaire is the result of a discussion between clinicians specialized in pediatric and obstetric anesthesia and researchers specialized in the neurocognitive development of children.

Several anamnestic data from the medical records of the patients and their child such as progress of pregnancy, childbirth history, history of general anesthesia during childhood, hospitalization during childhood,, will also be collected retrospectively on a standardized data collection sheet.

Statistical Methodology:

The number of subjects included in the Caen University Hospital cohort comprises : 31 patients in the "locoregional anesthesia" (LRA) group with a 1:2 matching with the "general anesthesia" (GA) group, resulting in 62 patients.

The "control" group is also matched with a 1:2 ratio with the "LRA" group, resulting in 62 patients.

The significance level is set at 5%. Data will be collected using Excel 2022 software (Microsoft Corporation, Redmond, WA, USA). Discrete variables will be expressed as number of cases (%). Continuous variables will be presented as mean ± standard deviations for normally distributed data or as median (95% confidence interval) for non-normally distributed data.

The statistical software used will be Statistica 12, Statsoft®.

Data Management:

The data will be entered into a spreadsheet for statistical analysis of the collected values. These data will only be used for this study, and the sponsor undertakes not to disclose them to third parties. The data processing will comply with the General Data Protection Regulation (GDPR) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Children born between 2011 and 2018 at Caen University Hospital
* Children whose mothers underwent surgery for non-obstetrical reasons under general or locoregional anesthesia, or did not undergo any surgical intervention.

Exclusion Criteria:

* Lost to follow-up
* Incomplete medical files
* Refusal of either parent or legal guardian
* Children with condition presenting independent risk factors for impaired neurocognitive development such as : neonatal hypoxia-ischemia, neurological disorder, neuromuscular disorder, complex cardiac or genetic disorders
* Children with a known or suspected genetic syndrome
* Preterm-born children (defined as birth at less than 37 weeks of amenorrhea)
* Cesarean-born children

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born between 2011 and 2018 at Caen University Hospital :
  * Whose mothers underwent general anesthesia for non-obstetric surgery during pregnancy (the "general anesthesia" group).
  * Whose mothers underwent locoregional anesthesia for non-obstetric surgery during pregnancy (the "locoregional anesthesia" group).
  * Whose mothers who did not undergo any surgical intervention during pregnancy (the "control" group).
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
The "Behavior Rating Inventory of Executive Function" composite score | Through the fourty minute phone call to the child's legal guardian. All phone calls will be conducted during the course of the study, which lasts an average of 2 months."
  The "Behaviour Rating Inventory of Executive Function" (BRIEF) is a parental questionnaire that assesses the executive functions of children aged 5 to 18 years old. It consists of 86 questions grouped into 8 scales: inhibition, flexibility, emotional control, initiation, material organization, working memory, planning/organization, and monitoring. It provides information on a global scale (score) regarding subtle and subclinical changes in various executive functions

SECONDARY OUTCOMES:
The child's cognitif functioning (at school, parental home, and during extracurricular activities), and medical history. | Through the fourty minute phone call to the child's legal guardian. All phone calls will be conducted the course during of the study, which lasts an average of 2 months."
  Progress of pregnancy, history of general anesthesia during childhood, hospitalization during childhood, non-febrile seizure during childhood, history of chronic otolaryngological pathology, specialized neuro-pediatric or child psychiatry follow-up, psychological or speech therapy in childhood, use of psychotropic medication, occasional psychological consultation, Psychological follow-up in childhood, speech therapy follow-up, diagnosed developmental disorder, reported school delay, school difficulties reported by teachers, specialized class or institution, experience of traumatic life events (bullying, death of a loved one), child's well-being in daily life: at school, at home, engagement in extracurricular activities and child's well-being, amount of screen time

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Salaün, MD PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- University Hospital Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salaun JP, Chagnot A, Cachia A, Poirel N, Datin-Dorriere V, Dujarrier C, Lemarchand E, Rolland M, Delalande L, Gressens P, Guillois B, Houde O, Levard D, Gakuba C, Moyon M, Naveau M, Orliac F, Orliaguet G, Hanouz JL, Agin V, Borst G, Vivien D. Consequences of General Anesthesia in Infancy on Behavior and Brain Structure. Anesth Analg. 2023 Feb 1;136(2):240-250. doi: 10.1213/ANE.0000000000006233. Epub 2022 Oct 27. PMID 36638508
- [Background] Bleeser T, Devroe S, Lucas N, Debels T, Van de Velde M, Lemiere J, Deprest J, Rex S. Neurodevelopmental outcomes after prenatal exposure to anaesthesia for maternal surgery: a propensity-score weighted bidirectional cohort study. Anaesthesia. 2023 Feb;78(2):159-169. doi: 10.1111/anae.15884. Epub 2022 Oct 25. PMID 36283123
- [Background] Shi Y, Hu D, Rodgers EL, Katusic SK, Gleich SJ, Hanson AC, Schroeder DR, Flick RP, Warner DO. Epidemiology of general anesthesia prior to age 3 in a population-based birth cohort. Paediatr Anaesth. 2018 Jun;28(6):513-519. doi: 10.1111/pan.13359. Epub 2018 Mar 13. PMID 29532559
- [Background] Marchesini V, Disma N. Anaesthetic neuroprotection in children: does it exist or is it all just bad? Curr Opin Anaesthesiol. 2019 Jun;32(3):363-369. doi: 10.1097/ACO.0000000000000723. PMID 30893117
- [Background] Paule MG, Li M, Allen RR, Liu F, Zou X, Hotchkiss C, Hanig JP, Patterson TA, Slikker W Jr, Wang C. Ketamine anesthesia during the first week of life can cause long-lasting cognitive deficits in rhesus monkeys. Neurotoxicol Teratol. 2011 Mar-Apr;33(2):220-30. doi: 10.1016/j.ntt.2011.01.001. Epub 2011 Jan 15. PMID 21241795
- [Background] Andropoulos DB, Greene MF. Anesthesia and Developing Brains - Implications of the FDA Warning. N Engl J Med. 2017 Mar 9;376(10):905-907. doi: 10.1056/NEJMp1700196. Epub 2017 Feb 8. No abstract available. PMID 28177852
- [Background] Walkden GJ, Gill H, Davies NM, Peters AE, Wright I, Pickering AE. Early Childhood General Anesthesia and Neurodevelopmental Outcomes in the Avon Longitudinal Study of Parents and Children Birth Cohort. Anesthesiology. 2020 Nov 1;133(5):1007-1020. doi: 10.1097/ALN.0000000000003522. PMID 32898216
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Warner DO, Zaccariello MJ, Katusic SK, Schroeder DR, Hanson AC, Schulte PJ, Buenvenida SL, Gleich SJ, Wilder RT, Sprung J, Hu D, Voigt RG, Paule MG, Chelonis JJ, Flick RP. Neuropsychological and Behavioral Outcomes after Exposure of Young Children to Procedures Requiring General Anesthesia: The Mayo Anesthesia Safety in Kids (MASK) Study. Anesthesiology. 2018 Jul;129(1):89-105. doi: 10.1097/ALN.0000000000002232. PMID 29672337
- [Background] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180
- [Background] McCann ME, de Graaff JC, Dorris L, Disma N, Withington D, Bell G, Grobler A, Stargatt R, Hunt RW, Sheppard SJ, Marmor J, Giribaldi G, Bellinger DC, Hartmann PL, Hardy P, Frawley G, Izzo F, von Ungern Sternberg BS, Lynn A, Wilton N, Mueller M, Polaner DM, Absalom AR, Szmuk P, Morton N, Berde C, Soriano S, Davidson AJ; GAS Consortium. Neurodevelopmental outcome at 5 years of age after general anaesthesia or awake-regional anaesthesia in infancy (GAS): an international, multicentre, randomised, controlled equivalence trial. Lancet. 2019 Feb 16;393(10172):664-677. doi: 10.1016/S0140-6736(18)32485-1. Epub 2019 Feb 14. PMID 30782342
- [Background] DiMaggio C, Sun LS, Li G. Early childhood exposure to anesthesia and risk of developmental and behavioral disorders in a sibling birth cohort. Anesth Analg. 2011 Nov;113(5):1143-51. doi: 10.1213/ANE.0b013e3182147f42. Epub 2011 Mar 17. PMID 21415431
- [Background] Zhang H, Du L, Du Z, Jiang H, Han D, Li Q. Association between childhood exposure to single general anesthesia and neurodevelopment: a systematic review and meta-analysis of cohort study. J Anesth. 2015 Oct;29(5):749-57. doi: 10.1007/s00540-015-2030-z. Epub 2015 May 23. PMID 26002228
- [Background] Clausen NG, Kahler S, Hansen TG. Systematic review of the neurocognitive outcomes used in studies of paediatric anaesthesia neurotoxicity. Br J Anaesth. 2018 Jun;120(6):1255-1273. doi: 10.1016/j.bja.2017.11.107. Epub 2018 Feb 3. PMID 29793593
- [Background] Walkden GJ, Pickering AE, Gill H. Assessing Long-term Neurodevelopmental Outcome Following General Anesthesia in Early Childhood: Challenges and Opportunities. Anesth Analg. 2019 Apr;128(4):681-694. doi: 10.1213/ANE.0000000000004052. PMID 30883414
- [Background] Yuki K, Matsunami E, Tazawa K, Wang W, DiNardo JA, Koutsogiannaki S. Pediatric Perioperative Stress Responses and Anesthesia. Transl Perioper Pain Med. 2017;2(1):1-12. PMID 28217718
- [Background] Wilder RT, Flick RP, Sprung J, Katusic SK, Barbaresi WJ, Mickelson C, Gleich SJ, Schroeder DR, Weaver AL, Warner DO. Early exposure to anesthesia and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Apr;110(4):796-804. doi: 10.1097/01.anes.0000344728.34332.5d. PMID 19293700
- [Background] Balinskaite V, Bottle A, Sodhi V, Rivers A, Bennett PR, Brett SJ, Aylin P. The Risk of Adverse Pregnancy Outcomes Following Nonobstetric Surgery During Pregnancy: Estimates From a Retrospective Cohort Study of 6.5 Million Pregnancies. Ann Surg. 2017 Aug;266(2):260-266. doi: 10.1097/SLA.0000000000001976. PMID 27617856
- [Background] Devroe S, Bleeser T, Van de Velde M, Verbrugge L, De Buck F, Deprest J, Devlieger R, Rex S. Anesthesia for non-obstetric surgery during pregnancy in a tertiary referral center: a 16-year retrospective, matched case-control, cohort study. Int J Obstet Anesth. 2019 Aug;39:74-81. doi: 10.1016/j.ijoa.2019.01.006. Epub 2019 Jan 12. PMID 30772120
- [Background] Vujic J, Marsoner K, Lipp-Pump AH, Klaritsch P, Mischinger HJ, Kornprat P. Non-obstetric surgery during pregnancy - an eleven-year retrospective analysis. BMC Pregnancy Childbirth. 2019 Oct 25;19(1):382. doi: 10.1186/s12884-019-2554-6. PMID 31653246
- [Background] Reitman E, Flood P. Anaesthetic considerations for non-obstetric surgery during pregnancy. Br J Anaesth. 2011 Dec;107 Suppl 1:i72-8. doi: 10.1093/bja/aer343. PMID 22156272
- [Background] Bleeser T, Van Der Veeken L, Fieuws S, Devroe S, Van de Velde M, Deprest J, Rex S. Effects of general anaesthesia during pregnancy on neurocognitive development of the fetus: a systematic review and meta-analysis. Br J Anaesth. 2021 Jun;126(6):1128-1140. doi: 10.1016/j.bja.2021.02.026. Epub 2021 Apr 6. PMID 33836853
- [Background] Zou S, Wei ZZ, Yue Y, Zheng H, Jiang MQ, Wu A. Desflurane and Surgery Exposure During Pregnancy Decrease Synaptic Integrity and Induce Functional Deficits in Juvenile Offspring Mice. Neurochem Res. 2020 Feb;45(2):418-427. doi: 10.1007/s11064-019-02932-z. Epub 2019 Dec 20. PMID 31858378
- [Background] Wu Z, Li X, Zhang Y, Tong D, Wang L, Zhao P. Effects of Sevoflurane Exposure During Mid-Pregnancy on Learning and Memory in Offspring Rats: Beneficial Effects of Maternal Exercise. Front Cell Neurosci. 2018 May 3;12:122. doi: 10.3389/fncel.2018.00122. eCollection 2018. PMID 29773978
- [Background] Dong C, Rovnaghi CR, Anand KJ. Ketamine exposure during embryogenesis inhibits cellular proliferation in rat fetal cortical neurogenic regions. Acta Anaesthesiol Scand. 2016 May;60(5):579-87. doi: 10.1111/aas.12689. Epub 2016 Jan 29. PMID 26822861
- [Background] Creeley CE, Dikranian KT, Dissen GA, Back SA, Olney JW, Brambrink AM. Isoflurane-induced apoptosis of neurons and oligodendrocytes in the fetal rhesus macaque brain. Anesthesiology. 2014 Mar;120(3):626-38. doi: 10.1097/ALN.0000000000000037. PMID 24158051
- [Background] Sprung J, Flick RP, Wilder RT, Katusic SK, Pike TL, Dingli M, Gleich SJ, Schroeder DR, Barbaresi WJ, Hanson AC, Warner DO. Anesthesia for cesarean delivery and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Aug;111(2):302-10. doi: 10.1097/ALN.0b013e3181adf481. PMID 19602960
- [Background] Robbins LS, Blanchard CT, Biasini FJ, Powell MF, Casey BM, Tita AT, Harper LM. General anesthesia for cesarean delivery and childhood neurodevelopmental and perinatal outcomes: a secondary analysis of a randomized controlled trial. Int J Obstet Anesth. 2021 Feb;45:34-40. doi: 10.1016/j.ijoa.2020.08.007. Epub 2020 Aug 25. PMID 33121885
- [Background] Ing C, Landau R, DeStephano D, Miles CH, von Ungern-Sternberg BS, Li G, Whitehouse AJO. Prenatal Exposure to General Anesthesia and Childhood Behavioral Deficit. Anesth Analg. 2021 Sep 1;133(3):595-605. doi: 10.1213/ANE.0000000000005389. PMID 33497062
- [Background] Baron IS. Behavior rating inventory of executive function. Child Neuropsychol. 2000 Sep;6(3):235-8. doi: 10.1076/chin.6.3.235.3152. No abstract available. PMID 11419452